CLINICAL TRIAL: NCT00757900
Title: Efficacy of Influenza Vaccine in HIV Infected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Shabir A Madhi, DST/NRF Vaccine Preventable Diseases (University of the Witwatersrand)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CHRU02 (Ethics ref no 080212)
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-09

CONDITIONS: HIV; Influenza; Vaccination; HIV Infections
Keywords: influenza, human
MeSH Terms: conditions — Influenza, Human; HIV Infections | interventions — mutagrip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): To receive a sub-unit influenza vaccine
  Interventions: Biological: MUTAGRIP
- 2 (No Intervention)

INTERVENTIONS:
Biological: MUTAGRIP — Purified polyvalent vaccine for active immunisation against influenza.The vaccine is an inactivated split virus mixture of different group A and B viral strains. One 0.5 ml dose, intramuscular route.
  Arms: 1

SUMMARY:
Vaccination of HIV infected individuals with the sub-unit influenza vaccine is safe; however it induces only moderate immune responses and likewise is modest in its protection compared to HIV uninfected individuals. Based upon the available data, the South African Thoracic Society has provisionally recommended the use of influenza vaccine in HIV infected individuals with CD4+ counts of > 200/ml and viral loads of < 100 000 copies/ml.(Green R et al. In press, SAMJ). This proposal is however based upon recommendations made elsewhere with minimal level of evidence regarding its benefit, and no evidence from countries with a high prevalence of HIV. Very few HIV infected adults, however, actually do receive influenza vaccine in South Africa, partly because of the absence of compelling data regarding the burden of disease in Africa as well as lack of vaccine effectiveness and issues related to physician awareness and access to influenza vaccine in the public immunization program.

The conflicting evidence, between developed countries and Africa, regarding the effectiveness of PPV highlight the drawbacks of extrapolating vaccine effectiveness data from developed countries to developing countries. Differences in the epidemiology of HIV between developed countries in which the prevalence of HIV is low to that of high-burden sub-Saharan African countries include:

* differences in the mode of transmission of HIV and demographics of the infected population.
* differences in standard of care, including access to prophylaxis against opportunistic infections and use of highly active anti-retroviral therapy (HAART)
* differences in risk for disease from opportunistic pathogens, e.g. Mycobacterium tuberculosis, etc.

These differences may all contribute to differences in the risk and severity of influenza illness among HIV infected adults from these communities as well as possibly responsiveness and effectiveness of vaccination.

The investigators are conducting a double-blinded, placebo controlled randomized trial at the HIV treatment clinic at Helen Joseph Hospital to determine the effectiveness of influenza vaccination in HIV infected adults in South Africa. The significance of the findings from this study will help quantify the burden of influenza illness in African HIV infected adults, as well as assist in making more informed recommendations for the use of influenza vaccine in HIV infected adults and in guiding national policy for preparing for a future influenza virus-pandemic.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected adult on stable first line HAART for more than 3 months or anti-retroviral naïve HIV infected adult with a CD4+ cell count >100 cells/ml performed within the previous 3 months in relation to the date of randomization.
* Age 18-55 years.
* Willing and able to maintain weekly contact at least during period of April - August (i.e. presupposed influenza period) either through SMS or telephonic contact.
* Willing and able to adhere to study protocol re: attendance to clinic for scheduled and illness visits.

Exclusion Criteria:

* Any contraindication to influenza vaccination, including known allergy to egg.
* Currently on treatment for tuberculosis or received treatment for tuberculosis in the past 6 months.
* History of chronic lung disease which required maintenance therapy either currently or in the past 6 months.
* Any contraindication to intramuscular injections.
* Current known grade 3 or grade 4 laboratory or clinical toxicity as per DAIDS toxicity tables.
* Any previous history of influenza or pneumococcal vaccination.
* Any plan to vaccinate against influenza or pneumococcal disease during the course of the study.
* Plan to emigrate from the study area within the next year.
* On steroid therapy for >21 days (current or within the past 30 days).
* In the investigators opinion unable to maintain study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 507 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
First episode of culture-confirmed influenza illness caused by community-acquired subtypes antigenically similar to the strains included in the influenza vaccine which occurred at least 14 days following study-vaccine administration. | 1st May 2008 and ending 30th September 2008.
The antibody response for each virus strain. Seroconversion will be defined as a ≥4-fold increase in antibody titer relative to that season's baseline titer for each strain.

SECONDARY OUTCOMES:
Incidence of solicited reactogenic events occurring within 72 hours of vaccination.
Changes in CD4+ cell count and HIV viral load.
Hospitalization or death for any physician-diagnosed respiratory illness in which influenza virus antigenically similar to vaccine strain is identified.

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MBBCH PhD, Principal Investigator — University of Witwatersrand, South Africa; Ian Sanne, MBBCh, Principal Investigator — Clinical HIV Research Unit
Locations (1):
- Helen Joseph Hospital, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Madhi SA, Maskew M, Koen A, Kuwanda L, Besselaar TG, Naidoo D, Cohen C, Valette M, Cutland CL, Sanne I. Trivalent inactivated influenza vaccine in African adults infected with human immunodeficient virus: double blind, randomized clinical trial of efficacy, immunogenicity, and safety. Clin Infect Dis. 2011 Jan 1;52(1):128-37. doi: 10.1093/cid/ciq004. PMID 21148531